CLINICAL TRIAL: NCT03654313
Title: A Phase 1 Randomized, Blinded, Placebo-controlled Study to Evaluate the Safety and Pharmacokinetics of Single and Multiple Ascending Doses of MEDI6570 in Subjects With Type 2 Diabetes Mellitus.
Brief Title: Single and Multiple Ascending Doses of MEDI6570 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4920C00001
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Atherosclerosis; Cardiovascular Disease
Keywords: Atherosclerosis; Cardiovascular Disease; CAD; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A MEDI6570 Cohort 1 (Experimental): Part A MEDI6570 Cohort 1 dose level
  Interventions: Biological: MEDI6570
- Part A MEDI6570 Cohort 2 (Experimental): Part A MEDI6570 Cohort 2 dose level
  Interventions: Biological: MEDI6570
- Part A MEDI6570 Cohort 3 (Experimental): Part A MEDI6570 Cohort 3 dose level
  Interventions: Biological: MEDI6570
- Part A MEDI6570 Cohort 4 (Experimental): Part A MEDI6570 Cohort 4 dose level
  Interventions: Biological: MEDI6570
- Part A Placebo (Placebo Comparator): Part A Placebo
  Interventions: Biological: Placebo
- Part B MEDI6570 Cohort 1 (Experimental): Part B MEDI6570 Cohort 1 dose level
  Interventions: Biological: MEDI6570
- Part B MEDI6570 Cohort 2 (Experimental): Part B MEDI6570 Cohort 2 dose level
  Interventions: Biological: MEDI6570
- Part B MEDI6570 Cohort 3 (Experimental): Part B MEDI6570 Cohort 3 dose level
  Interventions: Biological: MEDI6570
- Part B Placebo (Placebo Comparator): Part B Placebo
  Interventions: Biological: Part B Placebo
- Part A MEDI6570 Cohort 5 (Experimental): Part A MEDI6570 Cohort 5 Dose level
  Interventions: Biological: MEDI6570
- Part A MEDI6570 Cohort 6 (Experimental): Part A MEDI6570 Cohort 6 dose level
  Interventions: Biological: MEDI6570

INTERVENTIONS:
Biological: MEDI6570 — MEDI6570
  Arms: Part A MEDI6570 Cohort 1; Part A MEDI6570 Cohort 2; Part A MEDI6570 Cohort 3; Part A MEDI6570 Cohort 4; Part A MEDI6570 Cohort 5; Part A MEDI6570 Cohort 6; Part B MEDI6570 Cohort 1; Part B MEDI6570 Cohort 2; Part B MEDI6570 Cohort 3
Biological: Placebo — Placebo
  Arms: Part A Placebo
Biological: Part B Placebo — Placebo
  Arms: Part B Placebo

SUMMARY:
To evaluate the safety, tolerability, PK and immunogenicity of single and multiple ascending doses of MEDI6570 in subjects with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
A Phase 1 Randomized, Blinded, Placebo-controlled Study to Evaluate the Safety and Pharmacokinetics of Single and Multiple Ascending Doses of MEDI6570 in Subjects with Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria

* In Part A, subjects aged 18 through 65 inclusive at screening. In Part B, male subjects aged 18 through 65 inclusive, and female subjects aged 40 to 65 inclusive, at screening.
* Body mass index of 18 to 45 kg/m2.
* Subjects with T2DM on stable medical therapy for at least 6 weeks prior to screening with no clinically significant dose change and/or new medications in the recent 6 weeks
* Capable of giving written informed consent and adhere to visit/protocol schedule
* Female subjects must be of non-childbearing potential, confirmed at screening by one of the following: (a) Postmenopausal, defined as amenorrhea for ≥ 12 months following cessation of all exogenous hormonal treatments, and luteinizing hormone and follicle stimulating hormone (FSH) levels in the postmenopausal range. (b) Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy. Tubal ligation is not considered as irreversible surgical sterilization.
* Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide, and in addition the female partner must use 1 highly effective method of contraception.
* In Part B, subjects must meet CTA criteria as follows: (Estimated glomular filtration rate (eGFR) ≥ 60 mL/min/1.73m2. No allergy to iodinated contrast, no history of contrast induced nephropathy or no contraindication to beta blockers or nitroglycerin. No recent pulmonary embolism and must able to hold breath for at least 6 seconds. No history of coronary bypass surgery and no active arrhythmia on day of CTA scan (atrial fibrillation, atrial flutter, frequent premature atrial, or ventricular contractions).
* For Part A Cohort 6, subjects must be Japanese (eg, natives of Japan or Japanese Americans), defined as having both parents and four grandparents who are Japanese. This includes second and third generation subjects of Japanese descent whose parents or grandparents are living in a country other than Japan.

Exclusion Criteria

* History of any clinically important disease or disorder (not including T2DM) which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product, or planned surgical procedure before study completion.
* Female subjects who are pregnant and/or currently lactating.
* Any clinically important abnormalities in clinical chemistry, hematology, coagulation parameters, or urinalysis results -History of blood dyscrasia, hemostatic disorder, systemic bleeding, or prior trauma that places the subject at a higher risk of bleeding.
* History of vascular abnormalities including aneurysms, prior dissections; hx of severe hemorrhage, hematemesis, melena, haemoptysis, severe epistaxis, severe thrombocytopenia, intracranial hemorrhage, rectal bleeding, or major surgery/procedure within 3 months prior to Visit 1; a history suggestive of active peptic ulcer disease; or prior intracranial haemorrhage. -Dual-antiplatelet therapy, anticoagulation therapy or thrombolytic use, in the past month or planned use during the duration of the study. -Chronic aspirin therapy or chronic NSAID therapy.
* Clinically significant ECG that may interfere with the interpretation of serial ECG and QT interval changes screening. -Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or intraventricular conduction delay with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of ventricular hypertrophy or pre excitation. -Abnormal vital signs
* Hemoglobin A1c>9.0% measured at screening. HbA1c can be retested once after approximately 4 weeks.
* Clinically significant late diabetic complications including symptoms consistent with angina, congestive heart failure, and peripheral arterial disease (claudication), or other complications such as proliferative retinopathy, maculopathy, or gastroparesis.
* Any positive result at screening for serum hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV).
* History of cancer in the last 5 years, with the exception of non-melanoma skin cancer. -History of alcohol substance abuse within the past 6 months. A positive drug screen including recreational marijuana will be exclusionary. However, subjects with a documented medical need or prescription may be included at the discretion of the principal investigator.
* History of hypersensitivity or ongoing severe allergy or history of hypersensitivity to drugs with a similar chemical structure or calss to MEDI6570.
* History of ongoing infection or febrile illness within 30 days prior to Day 1.
* Current or previous use of systemic corticosteroids within 28 days prior to screening.
* Receipt of any investigational product or use of any biologics within 6 months or 5 half lives prior to screening (whichever is longer), or planned participation in an additional study of an investigational product therapy or biologic prior to end of follow up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and serious adverse events as a measure of safety and tolerability of MEDI6570 | Day 1 - Day 190 (Part A); Day 1 - Day 250 (Part B)
  Measured by the incidence of treatment- emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs)

SECONDARY OUTCOMES:
Pharmacokinetics of MEDI6570 AUC | Day 1 - Day 190 (Part A); Day 1 - Day 250 (Part B)
  Non-compartmental analysis will be performed for MEDI6570 treated subjects. Descriptive statistics for PK parameters will be provided
Pharmacokinetics of MEDI6570 Cmax | Day 1 - Day 190 (Part A); Day 1 - Day 250 (Part B)
  Non-compartmental analysis will be performed for MEDI6570 treated subjects. Descriptive statistics for PK parameters will be provided
Pharmacokinetics of MEDI6570 Tmax | Day 1 - Day 190 (Part A); Day 1 - Day 250 (Part B)
  Non-compartmental analysis will be performed for MEDI6570 treated subjects. Descriptive statistics for PK parameters will be provided
Pharmacokinetics of MEDI6570 Terminal Half life | Day 1 - Day 190 (Part A); Day 1 - Day 250 (Part B)
  Non-compartmental analysis will be performed for MEDI6570 treated subjects. Descriptive statistics for PK parameters will be provided
Immunogenicity rate | Day 1 - Day 190 (Part A); Day 1 - Day 250 (Part B)
  ADA incidence rate and titer will be tabulated for each treatment group. Samples confirmed positive for ADA will be tested and analyzed for nAB titer and summarized similarly.

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Sinsakul, Study Director — MedImmune LLC
Locations (9):
- United States (9):
  - Research Site, Anniston, Alabama
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, High Point, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Knoxville, Tennessee
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Vavere AL, Sinsakul M, Ongstad EL, Yang Y, Varma V, Jones C, Goodman J, Dubois VFS, Quartino AL, Karathanasis SK, Abuhatzira L, Collen A, Antoniades C, Koren MJ, Gupta R, George RT. Lectin-Like Oxidized Low-Density Lipoprotein Receptor 1 Inhibition in Type 2 Diabetes: Phase 1 Results. J Am Heart Assoc. 2023 Feb 7;12(3):e027540. doi: 10.1161/JAHA.122.027540. Epub 2023 Jan 23. PMID 36688371